CLINICAL TRIAL: NCT02496468
Title: The All Age Asthma Cohort (ALLIANCE) of the German Center for Lung Research (DZL), Pediatric Arm
Brief Title: Pediatric Arm of DZL All Age Asthma Cohort
Acronym: ALLIANCE
Status: Recruiting | Type: Observational
Sponsor: LMU Klinikum (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Center for Lung Research (Other); Comprehensive Pulmonary Center Munich (Unknown); Airway Research Center North (Unknown); Biomedical Research in Endstage and Obstructive Lung Disease Hannover (Unknown); Translational Lung Research Center Heidelberg (Unknown); Universities of Giessen and Marburg Lung Center (Unknown)
Responsible Party: Principal Investigator, Erika von Mutius, Prof. Dr. Bianca Schaub, LMU Klinikum
Other Study IDs: DZL_DA_AA-1
Record Dates: First submitted 2015-07-03; First posted 2015-07-14 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Asthma; Wheeze; Hypersensitivity; Endophenotype
Keywords: childhood asthma; preschool wheeze; adult asthma; transition; phenotype; endotype; trajectory
MeSH Terms: conditions — Asthma; Respiratory Sounds; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood (EDTA), serum, stool samples, whole blood cell pellets, primary nasal epithelial cells, induced sputum cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- new-onset wheeze/asthma: children with inhaled or systemic corticosteroid-/leukotriene receptor antagonist-naïve wheeze/asthma, will undergo follow-up after initial recruitment
- wheeze/asthma under controller therapy: children with wheeze/asthma, already under controller (inhaled or systemic corticosteroids or leukotriene receptor antagonist) therapy, will undergo follow-up after initial recruitment
- healthy controls: healthy age- and sex-matched controls, will not undergo follow-up after initial recruitment

SUMMARY:
Despite its common occurrence, still little is known about pathomechanisms determining different wheeze and asthma trajectories and phenotypes in children, and those beginning in adulthood. Therefore, deciphering underlying determinants for different childhood and adult asthma phenotypes is urgently needed to develop personalized treatment approaches targeting distinct underlying mechanisms. Thereby, secondary prevention early in the disease process can also be achieved. The decoding of such mechanisms and their translation to the individual patient is the aim of the Disease Area Asthma Allergy of the 'German Centre for Lung Research' (DZL).

DETAILED DESCRIPTION:
About 25-30% of children have at least one episode of wheeze before their 3rd birthday, but considerable clinical heterogeneity exists. Many of these children become symptom-free between 3 and 8 years of age, but some go on to persistent asthma in later childhood and adulthood. Despite its high prevalence, still little is known about pathomechanisms determining the different wheeze trajectories and phenotypes in children, and those beginning in adulthood. Frequency and severity of exacerbations may play an important role in the chronification process but underlying mechanisms are equally not well understood. Therefore, deciphering the role of airway mechanics, genetic, environmental and molecular determinants for different childhood and adult asthma phenotypes for exacerbations and chronification processes is urgently needed to develop personalized treatment approaches targeting distinct underlying mechanisms. Thereby, secondary prevention early in the disease process can also be achieved.

In order to do so, a clinical cohort for childhood asthma has been set up with identical, standardized instruments (quality assurance plan: standard operating procedures (SOPs) for clinical and lab modules, shipment, biobanking and analysis as well as quality control measures via audits and site visits have been developed) across the participating 'German Center for Lung Research' (DZL) sites. Here, new-onset steroid/leukotriene receptor antagonist (LTRA) naïve wheeze/asthma patients and wheeze/asthma patients under controller therapy are being recruited in addition to healthy controls. Following recruitment, regularly follow-ups and exacerbation visits of included patients are being performed with identical study instruments and meticulous quality control checks as at baseline.

PROJECT HYPOTHESES:

1. Specific molecular phenotypes are associated with distinct wheeze/asthma phenotypes and trajectories. Thereby, underlying mechanisms as well as predictors and biomarkers for persistent asthma will be identified.
2. Individuals at risk for exacerbations can be identified by clinical and molecular biomarkers, which will become novel targets for therapy and secondary prevention.

WORK PROGRAM:

Identification of molecular phenotypes, predictors and biomarkers for distinct wheeze/asthma phenotypes and trajectories.

The investigators aim to recruit over 1000 cases and controls to ensure sufficient statistical power for multivariate statistical analyses. Recruitment of study participants will be continued and cases will undergo 'deep phenotyping' as described below. In addition, healthy age and sex matched controls will be recruited. Cases and controls undergo a comprehensive clinical assessment including questionnaires (browser-based online data entry into extensive database with audit trail, plausibility and quality control checks implemented, data dictionary accessible), physical examination and lung function tests (spirometry and bodyplethysmography including bronchodilator response, multiple breath washout, exhaled nitric oxide). Biomaterials will be collected for analyses: i) blood samples; ii) nasal secretions; iii) pharyngeal swabs; iv) induced sputum; v) stool samples. Furthermore, epithelial cells will be collected by nasal brushings. Breath samples will be collected for analyses of volatile organic compounds. The cases will be followed up regularly using the same clinical tools and collecting the same biomaterials as at the initial visit to assess trajectories over time. Two closely interacting working groups have been established for all aims described: one lab and one data management/analysis group, each headed by expert members of the participating sites. The lab group will initiate and supervise all measurements of biomaterials; the data management/analysis group will expand the combined and shared data base and coordinate statistical analyses across sites. A common publication policy has already been developed. Using advanced bioinformatics, systems biology and machine learning approaches, the investigators will develop predictive (diagnostic) algorithms including clinical and molecular biomarkers for transient and persistent wheeze/asthma phenotypes and their trajectories. These analyses will also identify underlying mechanisms and thereby potential targets for future personalized therapy comparing childhood and adult findings. During data collection. The investigators attempt to minimize missing data. In all cases where missing data will reduce power for subsequent analyses, imputation will be used in order to omit power loss.

ELIGIBILITY:
Inclusion Criteria:

* informed consent by parents (and by children if age > 8 years)
* age 6 months to 18 years
* term delivery (≥ 37 weeks)
* active/passive understanding of German
* age 6 months - < 6 years: preschool wheeze (more than two episodes of wheeze during 12 months prior to inclusion)
* age at least 6 years: doctor diagnosed asthma (according to current guidelines)

Exclusion Criteria:

* known inborn or perinatal pulmonary disease
* airway malformation
* oxygen therapy after birth with a duration of more than 24 hours
* ventilator support or mechanical ventilation after birth
* diagnoses of cystic fibrosis; primary ciliary dyskinesia
* heart failure diagnosed after birth affecting pulmonary circulation
* major respiratory diseases such as e.g. interstitial lung disease
* any current non-atopic comorbidity
* fever of at least 38.5°C during the last two weeks prior to the planned first visit

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: preschool children with wheeze and school children as well as adolescents with asthma
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2013-01; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of asthma | At baseline and during yearly follow-ups up to 2 years
  Study participants will be assessed with regard to their development of asthma.
Prevalence of transient preschool wheeze | At baseline and during yearly follow-ups up to 2 years
  Study participants will be assessed with regard to their development of transient preschool wheeze.

SECONDARY OUTCOMES:
Prevalence of atopic sensitization | At baseline and during yearly follow-ups up to 2 years
  The prevalence of atopic sensitization will be measured by the detection of specific immunoglobin E against common aeroallergens.
Lung function | At baseline and during yearly follow-ups up to 2 years
  Study participants will be assessed with regard to lung function parameters (as measured by spirometry/bodyplethysmography and multiple-breath washouts (MBW)).
Levels of exhaled nitric oxide | At baseline and during yearly follow-ups up to 2 years
  Levels of exhaled nitric oxide (eNO) will be measured by chemoluminescence analyzers in combination with ultrasound-based flow measurement.
Frequency of acute exacerbations during previous 12 months | At baseline and during yearly follow-ups up to 2 years
  The frequency of acute exacerbations during previous 12 months will be assessed by questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Schaub, MD, Principal Investigator — Klinikum der Universitaet Muenchen, Comprehensive Pulmonary Center Munich; Gesine Hansen, MD, Principal Investigator — Biomedical Research in Endstage and Obstructive Lung Disease Hannover; Folke Brinkmann, MD, Principal Investigator — Airway Research Center North
Locations (5):
- Germany (5):
  - University Children's Hospital Cologne, Department of Paediatric Allergology and Pneumology, Cologne
  - Medizinische Hochschule Hannover, Biomedical Research in Endstage and Obstructive Lung Disease, Hanover
  - Universitaetsklinikum Schleswig-Holstein, Klinik für Kinder- und Jugendmedizin, Airway Research Center North, Lübeck
  - Klinik für Kinder- und Jugendmedizin, Universitaetsklinikum Giessen und Marburg GmbH, Universities of Giessen and Marburg Lung Center, Marburg
  - Klinikum der Universitaet Muenchen, Comprehensive Pulmonary Center Munich, Munich

REFERENCES:
- [Derived] Jakwerth CA, Weckmann M, Illi S, Charles H, Zissler UM, Oelsner M, Guerth F, Omony J, Nemani SSP, Grychtol R, Dittrich AM, Skevaki C, Foth S, Weber S, Alejandre Alcazar MA, van Koningsbruggen-Rietschel S, Brock R, Blau S, Hansen G, Bahmer T, Rabe KF, Brinkmann F, Kopp MV, Chaker AM, Schaub B, von Mutius E, Schmidt-Weber CB; ALLIANCE Study Group as part of the German Center for Lung Research. 17q21 Variants Disturb Mucosal Host Defense in Childhood Asthma. Am J Respir Crit Care Med. 2024 Apr 15;209(8):947-959. doi: 10.1164/rccm.202305-0934OC. PMID 38064241
- [Derived] Shahrokny P, Maison N, Riemann L, Ehrmann M, DeLuca D, Schuchardt S, Thiele D, Weckmann M, Dittrich AM, Schaub B, Brinkmann F, Hansen G, Kopp MV, von Mutius E, Rabe KF, Bahmer T, Hohlfeld JM, Grychtol R, Holz O. Increased breath naphthalene in children with asthma and wheeze of the All Age Asthma Cohort (ALLIANCE). J Breath Res. 2023 Oct 12;18(1). doi: 10.1088/1752-7163/acf23e. PMID 37604132
- [Derived] Maison N, Omony J, Illi S, Thiele D, Skevaki C, Dittrich AM, Bahmer T, Rabe KF, Weckmann M, Happle C, Schaub B, Meyer M, Foth S, Rietschel E, Renz H, Hansen G, Kopp MV, von Mutius E, Grychtol R; ALLIANCE Study Group; ALLIANCE Study Group; Fuchs O, Roesler B, Welchering N, Kohistani-Greif N, Kurz J, Landgraf-Rauf K, Laubhahn K, Liebl C, Ege M, Hose A, Zeitlmann E, Berbig M, Marzi C, Schauberger C, Zissler U, Schmidt-Weber C, Ricklefs I, Diekmann G, Liboschik L, Voigt G, Sultansei L, Nissen G, Konig IR, Kirsten AM, Pedersen F, Watz H, Waschki B, Herzmann C, Abdo M, Biller H, Gaede KI, Bovermann X, Steinmetz A, Husstedt BL, Nitsche C, Veith V, Szewczyk M, Brinkmann F, Malik A, Schwerk N, Dopfer C, Price M, Jirmo AC, Habener A, DeLuca DS, Gaedcke S, Liu B, Calveron MR, Weber S, Schildberg T, van Koningsbruggen-Rietschel S, Alcazar M. T2-high asthma phenotypes across lifespan. Eur Respir J. 2022 Sep 29;60(3):2102288. doi: 10.1183/13993003.02288-2021. Print 2022 Sep. PMID 35210326
- [Derived] Weckmann M, Bahmer T, Sand JM, Rank Ronnow S, Pech M, Vermeulen C, Faiz A, Leeming DJ, Karsdal MA, Lunding L, Oliver BGG, Wegmann M, Ulrich-Merzenich G, Juergens UR, Duhn J, Laumonnier Y, Danov O, Sewald K, Zissler U, Jonker M, Konig I, Hansen G, von Mutius E, Fuchs O, Dittrich AM, Schaub B, Happle C, Rabe KF, van de Berge M, Burgess JK, Kopp MV; ALLIANCE Study Group as part of the German Centre for Lung Research (DZL). COL4A3 is degraded in allergic asthma and degradation predicts response to anti-IgE therapy. Eur Respir J. 2021 Dec 9;58(6):2003969. doi: 10.1183/13993003.03969-2020. Print 2021 Dec. PMID 34326188
- [Derived] Skevaki C, Tafo P, Eiringhaus K, Timmesfeld N, Weckmann M, Happle C, Nelson PP, Maison N, Schaub B, Ricklefs I, Fuchs O, von Mutius E, Kopp MV, Renz H, Hansen G, Dittrich AM; ALLIANCE Study Group. Allergen extract- and component-based diagnostics in children of the ALLIANCE asthma cohort. Clin Exp Allergy. 2021 Oct;51(10):1331-1345. doi: 10.1111/cea.13964. Epub 2021 Jun 26. PMID 34128558
- [Derived] Fuchs O, Bahmer T, Weckmann M, Dittrich AM, Schaub B, Rosler B, Happle C, Brinkmann F, Ricklefs I, Konig IR, Watz H, Rabe KF, Kopp MV, Hansen G, von Mutius E; ALLIANCE Study Group as part of the German Centre for Lung Research (DZL). The all age asthma cohort (ALLIANCE) - from early beginnings to chronic disease: a longitudinal cohort study. BMC Pulm Med. 2018 Aug 20;18(1):140. doi: 10.1186/s12890-018-0705-6. PMID 30126401
- See also: Click here for more information about the German Center for Lung Research (DZL) — http://www.dzl.de/index.php/en/
- See also: Click here for more information about the Disease Area Asthma and Allergy (DA AA) as part of the German Center for Lung Research (DZL) — http://www.dzl.de/index.php/en/research/disease-areas/asthma-and-allergy